CLINICAL TRIAL: NCT00507611
Title: Sentinel Lymph Node Mapping and Biopsy For Predicting the Axillary Lymph Node Status After Completion of Preoperative Neoadjuvant Systemic Chemotherapy in Patients Who Had Biopsy-Proven Axillary Lymph Node Involvement at Initial Presentation
Brief Title: Axillary Lymph Node Status After Completion of Preoperative Neoadjuvant Systemic Chemotherapy in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Povoski (Other)
Responsible Party: Sponsor-Investigator, Stephen Povoski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-06077
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Invasive Breast Cancer
Keywords: breast; sentinel lymph node; node mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm (Other): Patients will undergo preoperative lymphoscintigraphy in the nuclear medicine department to access axillary and extra-axillary sites of localization. Intraoperatively, patients will also be injected with approximately 4 to 5 mL of 1% isosulfan blue dye (by intradermal, intraparenchymal, or subareolar route). Patients will undergo intraoperative identification and biopsy of all SLN candidates. A confirmatory axillary lymph node dissection will then be performed on all patients.
  Interventions: Procedure: Sentinel node mapping

INTERVENTIONS:
Procedure: Sentinel node mapping — Patients will undergo preoperative lymphoscintigraphy in the nuclear medicine department to access axillary and extra-axillary sites of localization. Intraoperatively, patients will also be injected with approximately 4 to 5 mL of 1% isosulfan blue dye (by intradermal, intraparenchymal, or subareolar route). Patients will undergo intraoperative identification and biopsy of all SLN candidates. A confirmatory axillary lymph node dissection will then be performed on all patients.
  Other Names: SLN mapping

SUMMARY:
The purpose of the present proposed clinical trial will be to assess the utility of SLN mapping and biopsy for predicting the final axillary status after completion of preoperative neoadjuvant systemic chemotherapy in patients who had biopsy-proven positive axillary lymph nodes at initial presentation

DETAILED DESCRIPTION:
Multiple retrospective reports have verified the overall utility of post-treatment sentinel lymph node (SLN) mapping and biopsy for assessing the final axillary lymph node status in breast cancer patients who have undergone preoperative neoadjuvant systemic chemotherapy. However, to date, only one report, in abstract form, currently exists within the literature which specifically assesses the utility of post-treatment SLN mapping and biopsy after completion of preoperative neoadjuvant systemic chemotherapy in patients with biopsy-proven positive axillary lymph nodes at initial presentation.

The purpose of the present proposed clinical trial will be to assess the utility of SLN mapping and biopsy for predicting the final axillary status after completion of preoperative neoadjuvant systemic chemotherapy in patients who had biopsy-proven positive axillary lymph nodes at initial presentation.

All eligible patients must have biopsy-proven invasive breast cancer and must also have biopsy-proven involvement of the axillary lymph nodes at initial presentation. Biopsy-proven involvement of the axillary lymph nodes at initial presentation will be based on fine needle aspiration (FNA) cytology, core/Tru-cut biopsy, or pre-treatment SLN biopsy. All eligible patients will have undergone preoperative neoadjuvant systemic chemotherapy.

After completion of preoperative neoadjuvant systemic chemotherapy and on the day of definitive breast cancer surgery, patients will be injected intradermally with approximately 400 microcuries of Tc-99m sulfur colloid. Patients will undergo preoperative lymphoscintigraphy in the nuclear medicine department to access axillary and extra-axillary sites of localization. Intraoperatively, patients will also be injected with approximately 4 to 5 mL of 1% isosulfan blue dye (by intradermal, intraparenchymal, or subareolar route). Patients will undergo intraoperative identification and biopsy of all SLN candidates. A confirmatory axillary lymph node dissection will then be performed on all patients.

The SLN mapping and biopsy procedure that we are proposing to perform on these breast cancer patients with known positive axillary lymph nodes at initial presentation will be done in an identical fashion to the SLN mapping and biopsy procedure that is currently performed as a routine and acceptable standard of care on every breast cancer patient with a clinically negative axilla at presentation.

The primary endpoints of this study would be address the success of identification of the SLN and the accuracy of the SLN mapping and biopsy procedure in women having undergone preoperative neoadjuvant systemic chemotherapy who had biopsy-proven involvement of their axillary lymph nodes at initial presentation. We would like to show that the proportion of women with false negative SLN biopsy results is less than 10%.

The study will require a minimum of 49 women with newly diagnosed breast cancer with biopsy-proven involvement of their axillary lymph nodes at initial presentation that have undergone preoperative neoadjuvant systemic chemotherapy. The study accrual time may take in the range of approximately 24 to 36 months to complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female and 18 years of age or older.
* Patients must have a clinical T1, T2, or T3 tumor size.
* Patients must have a histopathologic tissue diagnosis of breast cancer by a core-type of breast biopsy
* Patients must have had biopsy-proven involvement of the axillary lymph nodes at initial presentation based on fine needle aspiration (FNA) cytology, core/Tru-cut biopsy, or pre-treatment SLN biopsy that will require an axillary lymph node dissection to be performed at the time of the definitive breast cancer surgery.
* Patients will have had to undergone preoperative neoadjuvant systemic chemotherapy.
* Patients may be candidates for either lumpectomy or mastectomy.
* Patients may have a history of a previously treated metachronous contralateral breast cancer in the past.
* Patients may have synchronous bilateral breast cancer.

Exclusion Criteria:

* Patients must not be pregnant (The absence of pregnancy must be documented by any one of the following: negative serum pregnancy test, the history of surgical sterilization, or the absence of menstruation for at least six months prior to enrollment in the study)
* Patients may not have a history of previous treated ipsilateral breast cancer in the past.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
the proportion of women with successful identification of the SLN with a 95% confidence interval of not greater than 10%. | up to 36 months
the accuracy with a 95% confidence interval of not greater than 10%. | up to 36 months
Insure the proportion of women with false negative SLN results do not exceed 10% | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Povoski, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu